CLINICAL TRIAL: NCT05773183
Title: Exploring the Relationship Between Androgen Metabolism, Metabolic Disease and Skeletal Muscle Energy Balance in Men
Acronym: MMetdMH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Steroid Metabolism Analysis Core, University of Birmingham (Unknown); University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: MMetDMH
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-12

CONDITIONS: Hypogonadism, Male; Testosterone Deficiency; Prostate Cancer; Androgen Deficiency; Metabolic Disease; Metabolic Syndrome; Metabolic Disturbance; Obesity; Cardiovascular Diseases; NAFLD; Diabetes
Keywords: mechanism; mechanistic study
MeSH Terms: conditions — Eunuchism; Prostatic Neoplasms; Metabolic Diseases; Metabolic Syndrome; Obesity; Cardiovascular Diseases; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus | interventions — Testosterone; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Samples for targeted and non targeted metabolomics Saliva samples for targeted metabolomics Urine samples for targeted metabolomics Skeletal muscle samples for non targeted metabolomics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OBS1 [Observational Cohort 1]: 20 Eugonadal Healthy men 20 Men with Testosterone Deficiency not currently on Testosterone replacement therapy
- IC1 [Interventional Cohort 1]: 20 Men with Testosterone Deficiency progressed from OBS1 6 months post initiation of testosterone replacement therapy
  Interventions: Drug: Testosterone
- IC2 [Interventional Cohort 2]: 20 men with prostate cancer planned for GnRH analogue therapy
  Interventions: Drug: GnRH

INTERVENTIONS:
Drug: Testosterone — In OBS1 20 men will be started on Testosterone replacement therapy as per routine clinical practice. Data collection will occur prior initiating therapy, and 6 months post
  Groups: IC1 [Interventional Cohort 1]
Drug: GnRH — 20 men in OBS2 planned for GnRH analogue therapy will undergo data collection prior, and 3 months post initiation of GnRH analogue therapy
  Other Names: GnRH analogue
  Groups: IC2 [Interventional Cohort 2]

SUMMARY:
This study relates to men with hypogonadism, a condition describing a deficiency of androgens such as testosterone. Deficiency of these hormones occurs in men due to testicular (primary) or hypothalamic-pituitary (secondary) problems or may be observed in men undergoing androgen deprivation therapy for prostate cancer.

Testosterone plays an important role in male sexual development and health, but also plays a key role in metabolism and energy balance. Men with testosterone deficiency have higher rates of metabolic dysfunction. This results in conditions such as obesity, nonalcoholic fatty liver disease, diabetes, and cardiovascular disease. Studies have confirmed that treating testosterone deficiency with testosterone can reduce the risk of some of these adverse metabolic outcomes, however cardiovascular mortality remains higher than the general population. We know that testosterone deficiency therefore causes metabolic dysfunction. However, research to date has not established the precise mechanisms behind this.

In men with hypogonadism there is a loss of skeletal muscle bulk and function. Skeletal muscle is the site of many critical metabolic pathways; therefore it is likely that testosterone deficiency particularly impacts metabolic function at this site. Men with testosterone deficiency also have excess fat tissue, this can result in increased conversion of circulating hormones to a type of hormone which further suppresses production of testosterone. The mechanism of metabolic dysfunction in men with hypogonadism is therefore multifactorial.

The purpose of this study is to dissect the complex mechanisms linking obesity, androgens and metabolic function in men. Firstly, we will carry out a series of detailed metabolic studies in men with testosterone deficiency, compared to healthy age- and BMI-matched men. Secondly, we will perform repeat metabolic assessment of hypogonadal men 6 months after replacement of testosterone in order to understand the impact of androgen replacement on metabolism. Lastly, we will perform the same detailed metabolic assessment in men with prostate cancer before and after introduction of a drug which causes testosterone deficiency for therapeutic purposes.

DETAILED DESCRIPTION:
Male hypogonadism occurs due to a deficiency of androgens such as testosterone due to either primary (testicular) or secondary (hypothalamic pituitary) pathology. The incidence of testosterone deficiency is likely to increase with more cancer survivors, opiate use, increased awareness and thus diagnosis of testosterone deficiency. Hypogonadism in males is an independent risk factor for the development of metabolic syndrome and is associated with increased prevalence of insulin resistance, type two diabetes, non-alcoholic fatty liver disease, visceral adiposity, and cardiovascular disease.

The relationship between hypogonadism and metabolic dysfunction is bidirectional with secondary hypogonadism documented in a large proportion of men with obesity without a testicular or central cause of androgen deficiency. A vicious cycle exists whereby increased adipose tissue in men with obesity results in depleting circulating testosterone stores due to increased aromatisation of testosterone to oestrogen and suppression of gonadotrophin mediated testosterone secretion via negative feedback. This perpetuates visceral adiposity in men with pre-existing metabolic dysfunction.

The hormonal impact of visceral adiposity plays a role in aggravating metabolic disease in men with hypogonadism however the initial metabolic perturbation causing obesity and metabolic disease in these men has not been established. It is probable skeletal muscle dysfunction is a major player. Skeletal muscle is the primary site for glucose uptake and utilisation and houses critical metabolic pathways such as oxidative phosphorylation in mitochondria. Men with hypogonadism experience loss of skeletal muscle bulk and function. Research has previously demonstrated that pathologic alterations in androgen exposure result in mitochondrial dysfunction in females. Studies have also confirmed improvements in mitochondrial function include increased phosphorylation of AMPKα in men with diabetes and hypogonadotropic hypogonadism and in animal models increased expression of genes related to mitochondrial respiration enzymes following introduction of testosterone(12). These findings hint at a pivotal role for androgens in mitochondrial function and energy biogenesis in skeletal muscle. However, to date no mechanistic study has established the precise cellular mechanisms adversely modified by androgen deficiency in males.

Induction of hypogonadism or medical castration is a well-established therapeutic goal in men with recurrent or metastatic hormonally driven prostate cancer. This is typically achieved with androgen deprivation therapy either a GnRH analogue or androgen receptor blockade. Over half of men receiving ADT for treatment of prostate cancer experience metabolic syndrome. These men represent an excellent biological model for studying the association between hypogonadism and metabolic syndrome however research to date has focused on establishing the association but not the responsible mechanisms.

This study will establish the mechanism of metabolic dysfunction in males with androgen deficiency. Firstly a cohort of men with hypogonadism prior to testosterone replacement will undergo detailed metabolic phenotyping using multiple approaches including metabolomic data from skeletal muscle samples, and metabolic parameters using serum samples. This data will be compared to age and weight matched eugonadal healthy controls before and after testosterone replacement as per routine clinical care. The same detailed metabolic phenotyping will be performed on men with prostate cancer before and after therapeutic induction of hypogonadism.

Our study will provide an unparalleled understanding of the tissue- and sex-specific role of androgens as a driver of metabolic dysfunction. Anticipated disturbances in mitochondrial function and energy biogenesis in androgen excess and deficiency will advance scientific knowledge and create potential for developing future tissue specific mediators of metabolic dysfunction in males with hypogonadism.

ELIGIBILITY:
Inclusion Criteria [OBS1 & IC1]:

* Able to provide consent
* Ages 18 - 60 years
* BMI 20 - 35 kg / m2

Inclusion Criteria [IC2]:

* Able to provide consent
* Ages 40-85 years
* BMI 20 - 35 kg / m2

Exclusion Criteria [OBS1 & IC1]:

* Contraindication to testosterone replacement for patients with hypogonadism
* BMI <20 or > 35 kg / m2
* Age < 18 or > 60 years
* Diabetes Mellitus
* Confirmed ischaemic heart disease
* In patients with secondary hypogonadism co-existence of any untreated pituitary hormone deficiencies (ACTH, TSH, GH deficiency)
* Glucocorticoid use via any route within the last three months
* Current intake of drugs known to impact upon steroid or metabolic function or intake of such drugs during the six months preceding the planned recruitment

Exclusion Criteria [IC2]:

* Diabetes mellitus
* Confirmed ischaemic heart disease
* Any glucocorticoid therapy in the last 3 months (inhaled/transdermal/systemic)
* BMI <20 or >35
* Pre-existing hormonal pathology - primary testicular or pituitary pathology
* Age <40 or >85

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Study Population: Observational Cohort 1 (OBS1):
  * 20 eugonadal healthy volunteer controls
  * 20 hypogonadal men pre initiation of testosterone replacement therapy
  Interventional Cohort 1 (IC1):
  • 20 hypogonadal men 6 months post initiation of testosterone replacement therapy
  Interventional Cohort 2 (IC2):
  • 20 men with prostate cancer pre and 3 months post initiation of GnRH analogue therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-12 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
To compare differences in non-targeted serum and skeletal muscle metabolomics in men with hypogonadism compared to controls | 24 months
  Differences in non-targeted serum and skeletal muscle metabolomics in men with hypogonadism compared to controls
To compare differences in non-targeted serum and skeletal muscle metabolomics in men with hypogonadism pre and post testosterone replacement | 24 months
  Differences in non-targeted serum and skeletal muscle metabolomics in men
To compare differences in steroid metabolomics in men with prostate cancer pre- and post-androgen deprivation therapy (ADT) | 24 months
  Differences in steroid metabolomics in men with prostate cancer pre- and post-androgen deprivation therapy (ADT)

SECONDARY OUTCOMES:
To compare differences in steroid metabolomics in men with hypogonadism compared to controls | 24 months
  Differences in serum, urinary and salivary steroid metabolism
To compare differences in steroid metabolomics in men with hypogonadism pre and post testosterone replacement | 24 months
  Differences in serum, urinary and salivary steroid metabolism
To compare differences in steroid metabolomics in men with prostate cancer pre- and post-androgen deprivation therapy | 24 months
  Differences in serum, urinary and salivary steroid metabolism
To compare differences in metabolic phenotype in (i) hypogonadal men compared to healthy men (ii) hypogonadal men pre and post testosterone replacement therapy (iii) men with prostate cancer post initiation of Androgen Deprivation Therapy | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No